CLINICAL TRIAL: NCT00600834
Title: A Prospective Cohort Study Evaluating the Incidence of Nephrogenic Systemic Fibrosis in Patients With Stages 3 to 5 Chronic Kidney Disease Undergoing MRI With the Injection of ProHance
Brief Title: Evaluation of the Risk of NSF Following ProHance Injection in Patients With Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: Bracco Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: PH-106
Record Dates: First submitted 2008-01-15; First posted 2008-01-25 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-10

CONDITIONS: Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Fixed tissue samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: patients with moderate CKD (stage 3, according to the classification of CKD by the National Kidney Foundation, i.e., with eGFR comprised between 30 and 59 mL/min/1.73m2)
- 2: patients with severe CKD or kidney failure (stages 4 and 5, according to the classification of CKD by the National Kidney Foundation, i.e., with eGFR stably below 30 mL/min/1.73m2).

SUMMARY:
The objective of this long term study is to prospectively compare the incidence of NSF in two cohorts (Cohort 1- patients with moderate chronic kidney disease eGFR 30-59 and Cohort 2- patients with severe chronic kidney disease or kidney failure eGFR <30).

ELIGIBILITY:
Inclusion Criteria:

COHORT 1

* Is going to receive or has received PROHANCE injection during an MRI examination;
* Has CKD with eGFR stably comprised between 30 and 59 mL/min/1.73m2, as calculated from a SCr value obtained from the local laboratory within 24 hours prior to the PROHANCE injection.
* Provides written informed consent and is willing to comply with protocol requirements.

OR

COHORT 2

* Is going to receive or has received PROHANCE injection during an MRI examination;
* Has CKD with eGFR below 30 mL/min/1.73m2, as calculated from a SCr value obtained from the local laboratory within 24 hours prior to the PROHANCE injection.
* Provides written informed consent and is willing to comply with protocol requirements.

Exclusion Criteria:

COHORT 1

* Has received a GBCA within the past 12 months prior to inclusion in this study;
* Has unstable kidney function;
* Has any medical condition or other circumstances which would significantly decrease the chances of obtaining reliable data and achieving study objectives;
* Has ever been suspected of, or diagnosed with, NSF prior to the study-specific MRI;
* Is unable or unwilling to return for necessary office visits, to be examined by dermatologists or to undergo deep skin biopsy should development of NSF be suspected.

OR

COHORT 2

* Has received a GBCA within the past 12 months prior to inclusion in this study;
* Has any medical condition or other circumstances which would significantly decrease the chances of obtaining reliable data and achieving study objectives;
* Has ever been suspected of, or diagnosed with, NSF prior to the study-specific MRI;
* Is unable or unwilling to return for necessary office visits, to be examined by dermatologists or to undergo deep skin biopsy should development of NSF be suspected.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 1000 patients in 2 cohorts who are going to receive or have received PROHANCE during an MRI examination as part of their routine clinical management. The cohorts are defined as:
  COHORT 1-
  600 patients of any age, with moderate CKD (stage 3, i.e., with eGFR stably comprised between 30 and 59 mL/min/1.73m2);
  COHORT 2-
  400 patients of any age, with severe CKD or kidney failure (stages 4 and 5, i.e., with eGFR below 30 mL/min/1.73m2).
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2008-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
To estimate and compare the incidence of NSF in the two cohorts defined. The incidence is defined for each cohort as the number of cases of NSF observed during the follow-up time period over the total number of eligible patients. | 1, 3, 6, 12, 18 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Gianpaolo Pirovano, MD, Study Director — Bracco Diagnostics, Inc
Locations (1):
- Bracco Diagnostic Inc., Princeton, New Jersey, United States